CLINICAL TRIAL: NCT06499987
Title: Outcome of Resection Anastomosis and Long Term Stenting With Montgomery Tube Operations in Management of Grade 3 Benign Laryngotracheal Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Awatef Mahmoud Ahmed, assistant lecturer of otorhinolaryngology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-24-06-01MD
Record Dates: First submitted 2024-06-26; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Grade 3 Benign Laryngotracheal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resection anastomosis (Active Comparator): resection of the stenotic part of the trachea and then doing re anastomosis
  Interventions: Procedure: resection anastomosis
- long term stenting with Montgomery tube (Active Comparator): application of T shaped Montgomery tube for 6 months
  Interventions: Procedure: resection anastomosis

INTERVENTIONS:
Procedure: resection anastomosis — resection of stenotic part of trachea and reanastmosis
  Other Names: long term stenting with Montgomery tube

SUMMARY:
Laryngotracheal stenosis is a challenging problem in the field of laryngology. In the majority of patients, acquired stenosis of the larynx and trachea is due to accidental trauma, prolonged intubations, or tracheostomy. Congenital stenosis, caustic injury, and granulomatous diseases are also etiological factors in laryngotracheal stenosis (Grenier PA et al, 2009).

Tracheal stenosis can occur following tracheostomy or endotracheal intubation with inappropriate cuff pressure. It is due to pressure necrosis at the site of the cuff. Initially, there is inflammation of the damaged mucosa with increased secretion and secondary infection. Prolonged ischemia and secondary infection cause necrosis of the tracheal wall and exposure and sequestration of the cartilaginous rings. This damage results in the formation of granulation tissue and collapse of the tracheal wall (Satish Nair et al, 2014).

The tracheal stenosis is classified as simple, which is a soft, short segment web-like narrowing often limited to the mucosa only or complex stenosis, which is a hard, long-segment stricture with destruction of tracheal cartilages and fibrosis. Post tracheostomy stenosis occurs most commonly at the stoma site or less commonly at the site where the tip of the tube has impinged on the tracheal mucosa (Liu J et al, 2015).

The symptoms are generally insidious. Most arise 1 to 6 weeks after extubation, and early symptoms are often not recognized. The most common symptoms include shortness of breath, cough, recurrent pneumonia, wheezing, stridor, and cyanosis over time. Dyspnea is often the symptom until the tracheal diameter is 50% smaller than normal. When the tracheal diameter is 25% of its normal size, dyspnea and stridor may occur even at rest. These symptoms can be confused with other respiratory diseases (Rubikas R et al, 2014).

ELIGIBILITY:
Inclusion Criteria:

- patients who are diagnosed with layngotracheal stenosis either post tracheostomy or post intubation

Exclusion Criteria:

* The exclusion criteria will be patients who underwent laryngeal split and cartilaginous grafting; patients who underwent carinal resection; patients with incomplete records; and resection due to conditions other than post intubation tracheal stenosis (e.g., airway tumors, idiopathic stenosis, trauma, Wegener' granulomatosis and chronic relapsing polychondritis).

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
successful | 12 months
  release of respiratory distress

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

REFERENCES:
- [Background] Weksler B. Commentary: The role of gastroesophageal reflux in patients with acquired tracheal stenosis. J Thorac Cardiovasc Surg. 2019 Dec;158(6):1708-1709. doi: 10.1016/j.jtcvs.2019.08.071. Epub 2019 Sep 19. No abstract available. PMID 31604634
- [Background] Belafsky PC, Postma GN, Koufman JA. The validity and reliability of the reflux finding score (RFS). Laryngoscope. 2001 Aug;111(8):1313-7. doi: 10.1097/00005537-200108000-00001. PMID 11568561
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Liu J, Zhang CP, Li Y, Dong S. Post-intubation tracheal stenosis after management of complicated aortic dissection: a case series. J Cardiothorac Surg. 2015 Nov 4;10:148. doi: 10.1186/s13019-015-0357-z. PMID 26537875